CLINICAL TRIAL: NCT04891640
Title: Biologic Abatement and Capturing Kids' Outcomes and Flare Frequency in Juvenile Spondyloarthritis (BACK-OFF JSpA)
Brief Title: Biologic Abatement and Capturing Kids' Outcomes and Flare Frequency in Juvenile Spondyloarthritis
Acronym: BACK-OFF JSpA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21-018442; : GRT-00001036 (Other Grant/Funding Number: PCORI)
Record Dates: First submitted 2021-05-14; First posted 2021-05-18 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-08

CONDITIONS: Juvenile Spondyloarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- TNFi Standard Therapy (Active Comparator): Continue fixed standard treatment (i.e., no change from current therapy)
  Interventions: Other: Standard TNFi Therapy
- TNFi fixed longer dosing intervals (Experimental): Fixed longer dosing intervals of TNFi (i.e., increased time between doses)
  Interventions: Other: TNFi fixed longer dosing intervals
- TNFi Therapy Withdrawal (Experimental): Stop TNFi treatment
  Interventions: Other: Stop TNFi treatment

INTERVENTIONS:
Other: Standard TNFi Therapy — Participants randomly assigned to this arm will continue taking their TNFi medication as currently prescribed.
  Arms: TNFi Standard Therapy
Other: TNFi fixed longer dosing intervals — Participants randomly assigned to this arm will increase the time between TNFi medication doses.
  * Adalimumab- from every 2 to 3 weeks
  * Certolizumab- from every 2 to 4 weeks
  * Etanercept- from every 1 to 2 weeks
  * Golimumab- from every 4 to 6 weeks
  * Infliximab- from baseline to baseline + 2 weeks
  Arms: TNFi fixed longer dosing intervals
Other: Stop TNFi treatment — Participants randomly assigned to this arm will stop TNFi medication.
  Arms: TNFi Therapy Withdrawal

SUMMARY:
This randomized pragmatic trial will generate knowledge about strategies used to de-escalate tumor necrosis factor inhibitor (TNFi) therapy in patients with juvenile spondyloarthritis with sustained inactive disease and are treated at one of the 29 participating pediatric healthcare systems. This open label study will be conducted in the setting of routine clinical care and will compare the risk and timing of flare (Aim 1) and patients' lived experiences (Aim 2) across three arms.

DETAILED DESCRIPTION:
This project is a prospective, 12-month pragmatic randomized trial embedded within routine clinical care. Children with spondyloarthritis who have maintained inactive disease on a clinically prescribed standard dosing of a TNFi for 6 months or longer will be eligible for enrollment. Children will be randomized to one of the following alternative approaches: continued fixed standard dosing (arm 1), fixed longer dosing intervals of TNFi (arm 2), or stopping TNFi (arm 3). The recommended visit frequency is every 3 months through the study endpoint at 12 months. After subjects have followed their treatment assignment for 12 months, those who have not flared may modify their treatment regimen as per shared decision making between themselves and the treating physician. All participants will be monitored for 24 additional months for long-term outcomes after the intervention period.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females age 8 to 21 years
2. Juvenile SpA diagnosis (symptom onset before their 16th birthday):

   Pediatric Rheumatology International Trials Organization (PRINTO) revision of the The International League of Associations for Rheumatology (ILAR) criteria enthesitis/spondylitis-related Juvenile idiopathic arthritis (JIA)
   * Peripheral arthritis and enthesitis, or
   * Arthritis or enthesitis, plus ≥ 3 months of inflammatory back pain and sacroiliitis on imaging, or
   * Arthritis or enthesitis plus 2 of the following: (1) sacroiliac joint tenderness; (2) inflammatory back pain; (3) presence of Human leukocyte antigen (HLA-B27) ; (4) acute (symptomatic) anterior uveitis; and (5) history of a SpA in a first-degree relative
3. Currently taking one of the following TNFi therapies (Adalimumab, Certolizumab, Etanercept, Golimumab, Infliximab) at standard doses and dosing intervals
4. Have reached a clinically inactive disease state for a minimum of six months, as determined by treating physician
5. English speaking or Spanish speaking
6. Interested and willing to de-escalate TNFi therapy

Exclusion Criteria:

1) History of inflammatory bowel disease, history of uveitis that was not adequately controlled with localized ophthalmic treatment or psoriasis that pre-dates the start of TNFi therapy or psoriasis that started after TNFi therapy and has required more than topical therapy for control

Ages: 8 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 164 (Actual)
Dates: Start 2021-11-11 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Juvenile Spondyloarthritis (JSpA) flare | 12 months
  JSpA flare is defined as clinically meaningful worsening in ≥3 of the following: caregiver/patient assessment of well-being, physician assessment of disease activity, caregiver/patient assessment of pain, physical function, and active joint count. Meaningful change for well-being, disease activity, and pain are an increase of ≥2 on visual analogue scale (range 0-10 with higher scores indicating poorer well-being, higher disease activity, and higher magnitude of pain). Meaningful change in function is defined as ≥3 unit change in the PROMIS mobility or upper extremity T-scores. The Patient-Reported Outcomes Measurement Information System (PROMIS) short forms include 8 questions and a T-score of '50' represents the healthy population mean score with standard deviation of 10. Active joint count is defined as the number of joints with swelling or, in the absence of swelling, limitation of motion accompanied by pain or warmth as per the physician examination.

SECONDARY OUTCOMES:
Pain interference (as measured by the PROMIS short form) | 12 months
  Pain interference (as measured by the PROMIS short form) of children with spondyloarthritis in the three treatment arms. The PROMIS short form is a validated questionnaire that measures the self-reported consequences of pain on relevant aspects of a person's life.The PROMIS short form includes 8 questions and a T-score of '50' represents the healthy population mean score with standard deviation equal to 10.

CONTACTS AND LOCATIONS:
Locations (31):
- United States (30):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Phoenix Children's, Phoenix, Arizona
  - Children's Hospital Los Angeles, Los Angeles, California
  - Stanford University, Palo Alto, California
  - Children's Hospital of Colorado, Aurora, Colorado
  - Nemours Children's Hospital, Wilmington, Delaware
  - Children's National Health System, Washington D.C., District of Columbia
  - Nemours Children's Health, Orlando, Florida
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Riley Hospital for Children at IU Health, Indianapolis, Indiana
  - University of Iowa Stead Family Children's Hospital, Iowa City, Iowa
  - Boston Children's Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - University of Minnesota Masonic Children's Hospital, Minneapolis, Minnesota
  - Children's Mercy Hospital, Kansas City, Missouri
  - St. Louis Children's Hospital, St Louis, Missouri
  - Hospital for Special Surgery, New York, New York
  - Cohen Children's Medical Center, Queens, New York
  - Akron Children's Hospital, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Randall Children's Hospital at Legacy Emanuel, Portland, Oregon
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - UPMC Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Vanderbilt Children's Hospital, Nashville, Tennessee
  - UT Southwestern Medical Center, Dallas, Texas
  - Texas Children's Hospital - Baylor College of Medicine, Houston, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - Seattle Children's Hospital, Seattle, Washington
- The Hospital for Sick Children, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Weiss PF, Sears CE, Brandon TG, Forrest CB, Neu E, Kohlheim M, Leal J, Xiao R, Lovell D. Biologic Abatement and Capturing Kids' Outcomes and Flare Frequency in Juvenile Spondyloarthritis (BACK-OFF JSpA): study protocol for a randomized pragmatic trial. Trials. 2023 Feb 8;24(1):100. doi: 10.1186/s13063-022-07038-6. PMID 36755328